CLINICAL TRIAL: NCT06150352
Title: Exploring the Association Between Cognitive Function, Obstructive Sleep Apnea and Brain Imaging, and the Determinants of Neurocognitive Decline in Subjects With Subjective or Mild Cognitive Impairment
Brief Title: Sleep Apnea, Neurocognitive Decline and Brain Imaging in Patients With Subjective or Mild Cognitive Impairment
Status: Recruiting | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Mary Ip Sau-man, Emeritus Professor, The University of Hong Kong
Other Study IDs: UW 23-291
Record Dates: First submitted 2023-10-12; First posted 2023-11-29 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Obstructive Sleep Apnea; Mild Cognitive Impairment; Subjective Cognitive Impairment
Keywords: Obstructive sleep apnea; Neurocognitive function; CPAP
MeSH Terms: conditions — Sleep Apnea, Obstructive; Cognitive Dysfunction | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood for apolipoprotein E status
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Subjective or mild cognitive impairment patients: Subjective or mild cognitive impairment patients with or without CPAP treatment
  Interventions: Device: Continuous Positive Airway Pressure or other management for OSA per clinical indications.

INTERVENTIONS:
Device: Continuous Positive Airway Pressure or other management for OSA per clinical indications. — PAP therapy or other management will be advised for subjects with OSA per usual clinical criteria

SUMMARY:
Obstructive sleep apnea (OSA) is recurrent episodes of partial or complete obstruction of the upper airway during sleep that causes intermittent hypoxia and sleep fragmentation and potentially lead to cardiometabolic and neurocognitive sequelae. Chronic intermittent hypoxia, sleep fragmentation of OSA, and insufficient sleep have been significantly associated with higher risks of neurocognitive impairment, including mild cognitive impairment (MCI) and Alzheimer's disease. Thus, sleep and sleep apnea might be modifiable factors to neurocognitive impairment.

Positive airway pressure (PAP) is the first line of treatment to maintain open airways for patients with OSA. Improving sleep, sleep apnea and circadian function could be a high-value intervention target to alleviate cognitive impairment and decline in subjects with mild neurocognitive impairment.

Amyloid accumulation in brain tissue is a distinct feature of Alzheimers' disease, which is associated with potential impairment of neurocognition clinically. It predicts memory decline in initially cognitively unimpaired individuals.

The study explores the associations between sleep apnea, cognitive function and cerebral imaging and the role of PAP therapy on neurocognitive trajectory in these patients with subjective cognitive impairment /mild cognitive impairment (SCI/MCI).

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is recurrent episodes of partial or complete obstruction of the upper airway during sleep . Chronic intermittent hypoxia, sleep fragmentation of OSA, and insufficient sleep have been significantly associated with higher risks of neurocognitive impairment, including mild MCI and Alzheimer's disease. Thus, sleep and sleep apnea might be modifiable factors contributing towards neurocognitive impairment . Improving sleep and sleep apnea could be a high-value intervention to alleviate cognitive impairment and decline in subjects with mild neurocognitive impairment.

Amyloid accumulation in brain tissue is a distinct feature of Alzheimer's disease, which is associated with potential impairment of neurocognition clinically. It predicts memory decline in initially cognitively unimpaired individuals. Research suggested that cerebrospinal fluid amyloid-β42 levels showed significant differences in subjects with moderate/severe OSA compared with healthy control.

Investigators hypothesize that (i) OSA is a determinant of neurocognitive decline, and regular PAP therapy for OSA could reduce this decline in subjects presenting with subjective cognitive impairment (SCI) or MCI; (ii) OSA may contribute to cerebral amyloid burden in these subjects with clinical diagnosis of SCI/MCI.

This study (i) assesses the role of obstructive sleep apnea as a potential determinant of neurocognitive status and the impact of OSA therapy (CPAP or other interventions) on neurocognitive decline (ii) evaluates if OSA increases cerebral amyloid deposition using PET imaging.

Subjects are recruited from Memory clinic and who have undergone a study with sleep questionnaires, neurocognitive tests and home sleep apnea test (HSAT). Subjects with OSA (identified on HSAT) will be referred for management of OSA per usual clinical criteria. Sleep questionnaires and cognitive assessment tests will be reassessed at six months, one year, two year and 3 year, and determinants to neurocognitive changes will be analyzed.

Amyloid PET-MRI brain will also be done at baseline. Owing to resource constraints, investigators can only provide PET-MRI investigation for 90 subjects ( 60 subjects with moderate/severe OSA to be compared with 30 subjects with no/mild OSA) .

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 - 80 years
* Diagnosis of mild cognitive impairment based on Peterson's criteria.
* Diagnosis of subjective cognitive impairment, based on the subjective complaint of cognitive impairment, but with an unremarkable assessment of the Hong Kong version of Montreal cognitive Assessment scores
* Able to speak and read Chinese
* Adequate visual and auditory to perform a cognitive test
* Subjects with moderate-severe OSA or No OSA (diagnosis based on sleep study) would be invited for baseline PET-MRI brain scan

Exclusion Criteria:

* Diagnosed psychiatric illness with or without medication, e.g. major depressive disorder.
* Other clear organic causes of cognitive impairment, e.g. vascular cognitive impairment, brain tumour, dementia with Lewy body, mild cognitive impairment with Lewy body, Parkinson's disease, normal pressure hydrocephalus, neurosyphilis, autoimmune encephalitis, substance abuse, history of alcohol abuse.
* Diagnosis of cancer on active treatment
* Contraindications to PET-CT or MRI brain scan (excluded for neuroimaging studies)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruit in the Memory clinic or Sleep clinic, Queen Mary Hospital
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2023-09-26 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in neurocognitive function (ADAS Cog) | Baseline, 6 months, 1 year, 2 year, 3 year
  Measured by ADAS-Cog. The scores range from 0 to 70, "0" is the best possible score and "70" is the worst possible score.
Cerebral amyloid update in moderate to severe OSA and no to mild OSA | Baseline
  The brain images for each subject will consist of fused MRI (3D MPRAGE) and 18F-Flutemetamol PET images. The scans were visually interpreted as positive (abnormal) or negative (normal) by a trained neuroradiologist based on uptake of 18F-Flutemetamol.

SECONDARY OUTCOMES:
Change in ability to inhibit cognitive interference | Baseline, 6 months, 1 year, 2 year, 3 year
  Measured by Stroop Colour and Word Test (SCWT). Scored by time and error. A longer time indicates a worst score, while a shorter time indicates a better score.
Change in neurocognitive function (MoCA) | Baseline, 6 months, 1 year, 2 year, 3 year
  Measured by Montreal Cognitive Assessment (MoCA) score. The scores range from 0 to 30, "0" is the worst possible score and "30" is the best possible score.
Change in sleep profile and quality | Baseline, 6 months, 1 year, 2 year, 3 year
  Measured by Severe Insomnia Index. Each item asks the individual to rate the severity of his or her symptoms with a 4-point Likert scale. The total score ranges from 0 to 28. The higher the scores the greater the severity of insomnia
Change in sleep apnea symptoms | Baseline, 6 months, 1 year, 2 year, 3 year
  Measured by Pittsburgh Sleep Quality Index. Each of the sleep components yields a score ranging from 0 to 3, with 3 indicating the greatest dysfunction. The sleep component scores are summed to yield a total score ranging from 0 to 21, with the higher total score indicating worse sleep quality.
Change in daytime sleepiness | Baseline, 6 months, 1 year, 2 year, 3 year
  Measured by Epworth Sleepiness Scale. Each item asks the individual to rate their daytime sleepiness. The total score ranges from 0 to 24. The higher the scores, the greater the severity of daytime sleepiness
Change in insomnia symptoms | Baseline, 6 months, 1 year, 2 year, 3 year
  Measured by Severe Insomnia Index. Each item asks the individual to rate the severity of his or her symptoms with a 4-point Likert scale. The total score ranges from 0 to 28. The higher the scores, the greater the severity of insomnia
Change in depression symptoms | Baseline, 6 months, 1 year, 2 year, 3 year
  Measured by Geriatric Depression Scale - short form. The score ranges from 0 to 15. The higher the scores the more severe of depression.
Neuroimaging outcomes between two groups of subjects with moderate-severe OSA or no-mild OSA | Baseline
  A. Cerebral amyloid burden as measured by SUVR global and regional scores on 18F-Flutemetamol PET-CT imaging:
  Normalized for injected dose and body weight of each subject, standardized uptake values (SUVs) are calculated in 16 Alzheimer's disease signature brain regions by Cortex-ID softward (General Electric Healthcare Ltd., USA). The composite SUVR representing the global amyloid burden is the average SUVR value of the area-weighted mean for the 16 cortical ROIs;
  B. Cortical brain volumes based on brain segmentation using 3D T1-MPRAGE images by Freesurfer software, including total, deep gray and hippocampal volumes; temporal, parietal, frontal and occipital cortical volumes; and Alzheimer's signature regional volumes

CONTACTS AND LOCATIONS:
Overall Officials: Mary SM Ip, MD, Principal Investigator — School of Clinical Medicine, The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bao YW, Chau ACM, Chiu PK, Shea YF, Kwan JSK, Chan FHW, Mak HK. Heterogeneity of Amyloid Binding in Cognitively Impaired Patients Consecutively Recruited from a Memory Clinic: Evaluating the Utility of Quantitative 18F-Flutemetamol PET-CT in Discrimination of Mild Cognitive Impairment from Alzheimer's Disease and Other Dementias. J Alzheimers Dis. 2021;79(2):819-832. doi: 10.3233/JAD-200890. PMID 33361593
- [Background] Collij LE, Mastenbroek SE, Salvado G, Wink AM, Visser PJ, Barkhof F, van Berckel BNM, Lopes Alves I. Regional amyloid accumulation predicts memory decline in initially cognitively unimpaired individuals. Alzheimers Dement (Amst). 2021 Aug 2;13(1):e12216. doi: 10.1002/dad2.12216. eCollection 2021. PMID 34368416
- [Background] Cui W, Duan Z, Li Z, Feng J. Assessment of Alzheimer's disease-related biomarkers in patients with obstructive sleep apnea: A systematic review and meta-analysis. Front Aging Neurosci. 2022 Oct 13;14:902408. doi: 10.3389/fnagi.2022.902408. eCollection 2022. PMID 36313031
- [Background] Emamian F, Khazaie H, Tahmasian M, Leschziner GD, Morrell MJ, Hsiung GY, Rosenzweig I, Sepehry AA. The Association Between Obstructive Sleep Apnea and Alzheimer's Disease: A Meta-Analysis Perspective. Front Aging Neurosci. 2016 Apr 12;8:78. doi: 10.3389/fnagi.2016.00078. eCollection 2016. PMID 27148046
- [Background] Jackson ML, Cavuoto M, Schembri R, Dore V, Villemagne VL, Barnes M, O'Donoghue FJ, Rowe CC, Robinson SR. Severe Obstructive Sleep Apnea Is Associated with Higher Brain Amyloid Burden: A Preliminary PET Imaging Study. J Alzheimers Dis. 2020;78(2):611-617. doi: 10.3233/JAD-200571. PMID 33016907
- [Background] Leng Y, McEvoy CT, Allen IE, Yaffe K. Association of Sleep-Disordered Breathing With Cognitive Function and Risk of Cognitive Impairment: A Systematic Review and Meta-analysis. JAMA Neurol. 2017 Oct 1;74(10):1237-1245. doi: 10.1001/jamaneurol.2017.2180. PMID 28846764
- [Background] Lutsey PL, Norby FL, Gottesman RF, Mosley T, MacLehose RF, Punjabi NM, Shahar E, Jack CR Jr, Alonso A. Sleep Apnea, Sleep Duration and Brain MRI Markers of Cerebral Vascular Disease and Alzheimer's Disease: The Atherosclerosis Risk in Communities Study (ARIC). PLoS One. 2016 Jul 14;11(7):e0158758. doi: 10.1371/journal.pone.0158758. eCollection 2016. PMID 27415826
- [Background] Buckley CJ, Sherwin PF, Smith AP, Wolber J, Weick SM, Brooks DJ. Validation of an electronic image reader training programme for interpretation of [18F]flutemetamol beta-amyloid PET brain images. Nucl Med Commun. 2017 Mar;38(3):234-241. doi: 10.1097/MNM.0000000000000633. PMID 27984539